CLINICAL TRIAL: NCT02462772
Title: Phase II Trial to Assess the Safety and Acceptability of the Long-acting Injectable HIV Integrase Inhibitor, Cabotegravir (GSK1265744), in HIV Uninfected Women in KwaZulu-Natal, South Africa
Brief Title: Safety and Acceptability of Cabotegravir in HIV Uninfected Women in KwaZulu-Natal, South Africa
Acronym: CAPRISA014
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for the AIDS Programme of Research in South Africa (Network)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Dr Salim S Abdool Karim, Principal Investigator, Centre for the AIDS Programme of Research in South Africa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CAPRISA 014
Record Dates: First submitted 2015-05-27; First posted 2015-06-04 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Human Immunodeficiency Virus
Keywords: Cabotegravir; safety; long-acting injectable; HIV prevention; acceptability
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — cabotegravir

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabotegravir (Experimental): Women randomised to the cabotegravir arm will receive daily oral cabotegravir (30 mg tablets) for approximately 30 days and thereafter will receive intra-muscular gluteal injections of cabotegravir LA (800 mg, administered as two 400 mg injections) every 12 weeks
  Interventions: Drug: cabotegravir
- Placebo (Placebo Comparator): Women randomised to the placebo arm will receive daily oral tablets (30 mg tablets) for approximately 30 days and thereafter will receive intra-muscular gluteal injections of Intralipid® 20% every 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: cabotegravir — Cabotegravir 30 mg tablets are formulated as white to almost white oval-shaped coated tablets for oral administration. The cabotegravir LA is formulated as a sterile white to slightly coloured suspension containing 400mg/2mL of cabotegravir LA for administration by IM injection.
  Other Names: GSK1265744
  Arms: Cabotegravir
Drug: Placebo — Placebo tablets for cabotegravir are formulated as white to almost white oval-shaped coated tablets to visually match the active cabotegravir tablets. Placebo for cabotegravir injectable suspension is Intralipid® 20%. Intralipid® is a fat emulsion with no pharmacological action. It is a white, milky emulsion, consisting of purified soyabean oil, purified egg phospholipids and anhydrous glycerol. Intralipid® 20% is supplied in infusion bags.
  Other Names: Intralipid® 20%
  Arms: Placebo

SUMMARY:
The CAPRISA 014 trial aims to assess the safety and acceptability of the long-acting (LA) injectable antiretroviral agent, cabotegravir LA (GSK1265744), in HIV uninfected women in KwaZulu-Natal, South Africa.

DETAILED DESCRIPTION:
The CAPRISA 014 trial is designed to establish the safety and acceptability of cabotegravir LA in sexually active, at-risk HIV-uninfected women. A total of 632 HIV uninfected women (18 to 30 years) from two sites in KwaZulu-Natal, South Africa will be enrolled. The trial will be approximately 24 months, with an additional 12 months post-trial safety observation. The study is divided into three periods:

Period 1 - Clinical trial oral lead-in (up to 34 days) - Consenting participants will be randomized to receive daily oral cabotegravir (30mg tablets) or daily oral placebo for approximately 30 days, to assess safety and tolerability prior to exposure to the LA injectable formulation.

Period 2 - Clinical trial follow-up with injectable (approximately 48-96 weeks) - Participants who have successfully completed Period 1 will receive intra-muscular (IM) gluteal injections of cabotegravir LA (800 mg, administered as two 400 mg injections) or placebo every 12 weeks. The end of Period 2 marks the completion of clinical trial follow-up.

Period 3 - Post-trial safety follow-up off-product (approximately 12 months) - During this post-trial safety observation period, participants will be followed up (off product) for approximately 12 months after completion of period 2.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent to be screened for, and to enrol in, the study.
* Able and willing to provide adequate locator information for study retention purposes.
* Sexually active, defined as having had vaginal intercourse at least once in the past 30 days prior to screening.
* HIV negative on testing performed by study staff
* Have a negative pregnancy test performed by study staff
* Agree to use a non-barrier form of contraceptive
* Agree to adhere to study visits and procedures.
* Haemoglobin > 11 g/dL,
* ALT < ULN
* AST < ULN
* Total bilirubin < Grade 1
* Direct bilirubin < ULN
* Creatinine clearance ≥60 mL/min
* Hepatitis B surface antigen (HBsAg) negative
* Hepatitis C Ab negative
* In general good health, as assessed clinically

Exclusion Criteria:

* Past or current participation in any other HIV interventional research study or other concurrent studies which may interfere with this study.
* Clinically significant cardiovascular disease, including:
* ECG with:
* heart rate <50 or >100 beats per minute (one repeat ECG is allowed during screening; can be performed on the same day)
* QRS duration >120 msec
* QTc interval (B or F) > 450 msec
* evidence of previous myocardial infarction (pathologic Q waves, S-T segment changes (except early repolarization)
* any conduction abnormality (including but not specific to left or right complete bundle branch block, Atrioventricular block [2nd degree (type II) or higher], Wolf Parkinson White syndrome)
* sinus pauses > 3 seconds
* any significant arrhythmia which, in the opinion of the Principal Investigator or designee, will interfere with the safety for the individual participant
* history of non-sustained (3 consecutive ventricular ectopic beats on ECG at screening or entry) or sustained ventricular tachycardia
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting surgery or percutaneous transluminal coronary angioplasty or any clinically significant cardiac disease
* Underlying skin disease or currently active skin disorder (e.g., infection, inflammation, dermatitis, eczema, psoriasis, urticaria). Mild cases of localized disease or other mild skin condition may not be exclusionary at the discretion of the Principal Investigator or designee.
* Has a tattoo or other dermatological condition overlying the buttock region which in the opinion of the Principal Investigator or designee, may interfere with interpretation of injection site reactions.
* History of acute or chronic liver disease (e.g., non-alcoholic or alcoholic steatohepatitis) or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome, asymptomatic gallstones, or cholecystectomy).
* Coagulopathy (primary or iatrogenic) which would contraindicate IM injection.
* Active or planned use of prohibited medications as described in the SSP manual (updated regularly from the Investigator's Brochure).
* Pregnant or currently breastfeeding, or intends to become pregnant and/or breastfeed during the study.
* Known Hypersensitivity to egg, soya or peanut protein.
* Has any other condition that, based on the opinion of the Principal Investigator or designee, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 36 months
  The incidence of increase in graded AEs and in particular liver enzymes (AST/ALT) at the level of Grade 3 or higher.

SECONDARY OUTCOMES:
Acceptability of study injections and oral tablets | 24 months
  Participant's opinions on the injections and tablets will be obtained through structured interviews.
Incidence of sexually transmitted infections | 36 months
  Incidence of HIV, HSV-2, HPV, gonorrhoea, chlamydia and trichomonas infections in women
Area under the plasma concentration versus time curve (AUC) of cabotegravir | 36 months
  Cabotegravir concentrations will be measured throughout the study
Impact on pregnancy | 36 months
  The incidence of pregnancy and pregnancy outcomes in women assigned to cabotegravir and placebo will be compared
Resistance to antiretroviral drugs | 36 months
  Viruses from HIV seroconverters will be sequenced and assessed for resistance mutations
HIV viral load in women who acquire HIV | 36 months
  HIV viral load (copies/ml) will be measured and compared between the cabotegravir and placebo arms

OTHER OUTCOMES:
Pharmacogenomics of cabotegravir | 36 months
  The impact of genetic polymorphisms on response to cabotagravir LA will be assessed
Impact of contraception on area under the plasma concentration versus time curve (AUC) of cabotegravir | 36 months
  Cabotegravir concentrations in women on DMPA will be compared to women on other forms of contraception

CONTACTS AND LOCATIONS:
Overall Officials: Salim S Abdool Karim, MBCHB, PhD, Principal Investigator — Centre for the AIDS Programme of Research in South Africa; Quarraisha Abdool Karim, PhD, Principal Investigator — Centre for the AIDS Programme of Research in South Africa; Leila E Mansoor, PhD, Principal Investigator — Centre for the AIDS Programme of Research in South Africa
Locations (2):
- South Africa (2):
  - CAPRISA eThekwini Research Clinic, Durban, KwaZulu-Natal
  - CAPRISA Vulindlela Research Clinic, eMafakatini, KwaZulu-Natal

REFERENCES:
- [Background] Radzio J, Spreen W, Yueh YL, Mitchell J, Jenkins L, Garcia-Lerma JG, Heneine W. The long-acting integrase inhibitor GSK744 protects macaques from repeated intravaginal SHIV challenge. Sci Transl Med. 2015 Jan 14;7(270):270ra5. doi: 10.1126/scitranslmed.3010297. PMID 25589631
- [Background] Spreen WR, Margolis DA, Pottage JC Jr. Long-acting injectable antiretrovirals for HIV treatment and prevention. Curr Opin HIV AIDS. 2013 Nov;8(6):565-71. doi: 10.1097/COH.0000000000000002. PMID 24100877